CLINICAL TRIAL: NCT03045263
Title: Pivotal Response Treatment Telemedicine
Brief Title: Pivotal Response Treatment (PRT) Telemedicine
Acronym: PRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1504015664
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pivotal Response Treatment (Active Comparator): Pivotal Response Training with children ages 3-6 years of age with an Autism Spectrum Disorder diagnosis
  Interventions: Behavioral: Pivotal Response Treatment
- Waitlist Control (No Intervention): Children in WL will be offered treatment following WL condition.

INTERVENTIONS:
Behavioral: Pivotal Response Treatment — Behavioral intervention for autism
  Other Names: PRT
  Arms: Pivotal Response Treatment

SUMMARY:
The purpose of this study is to evaluate the application of a modified version of PRT designed specifically as a parent-training model via telemedicine, with the goal of increasing access to empirically validated care. The project will feature an 18-week trial of parent training PRT via telemedicine in 12 cognitively able 3- to 6-year-old children with ASD. Intervention will focus on enhancing the following developmental skills: expressive and receptive language, play, and social interaction. Outcome measures will address changes in the aforementioned domains during structured observation and standardized assessment.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the application of a modified version of PRT designed specifically as a parent-training model via telemedicine, with the goal of increasing access to empirically validated care. The project will feature an 18-week trial of parent training PRT via telemedicine in 12 cognitively able 3- to 6-year-old children with ASD. Intervention will focus on enhancing the following developmental skills: expressive and receptive language, play, and social interaction. Outcome measures will address changes in the aforementioned domains during structured observation and standardized assessment.

ELIGIBILITY:
Inclusion Criteria:

* Fits age requirement: age 3-6 years
* Have been diagnosed previously with ASD and meet criteria for ASD when characterized by research team.
* be in good medical health
* be cooperative with testing
* english is a language spoken in the family
* full scale IQ > 70

Exclusion Criteria:

* significant hearing loss or other severe sensory impairment
* a fragile health status
* a history of significant head trauma or serious brain or psychiatric illness

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Behavioural Intervention Rating Scale (BIRS) | 10 weeks

SECONDARY OUTCOMES:
Client Credibility Questionnaire (CCQ) | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States